CLINICAL TRIAL: NCT01552850
Title: An Open-Label, Single-Dose, Randomized, Crossover Pharmacokinetics And Relative Bioavailability Study Of Three Modified 40 Mg Oxycodone Formulations Compared With 40 Mg Pf-00345439 Capsule Formulation In Healthy Volunteers
Brief Title: Pharmacokinetics And Relative Bioavailability Study Of Oxycodone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pain Therapeutics (Industry)
Responsible Party: Sponsor
Organization: PainT (Unknown)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B4501010
Record Dates: First submitted 2012-03-09; First posted 2012-03-13 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Pain
Keywords: pharmacokinetics; relative bioavailability; oxycodone
MeSH Terms: conditions — Pain | interventions — Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Oxycodone Formulation A Capsule (Experimental): single dose of 40 mg PF-00345439 capsule under 50 mg naltrexone block
  Interventions: Drug: Oxycodone
- Oxycodone Formulation B Capsule (Experimental): single dose of 40 mg PF-00345439 capsule under 50 mg naltrexone block
  Interventions: Drug: Oxycodone
- Oxycodone Formulation C Capsule (Experimental): single dose of 40 mg PF-00345439 capsule under 50 mg naltrexone block
  Interventions: Drug: Oxycodone
- Oxycodone Formulation D Capsule (Experimental): single dose of 40 mg PF-00345439 capsule under 50 mg naltrexone block
  Interventions: Drug: Oxycodone
- Oxycodone Oral Solution (Experimental): 40 mg oxycodone oral solution (5 mg/5 ml) under 50 mg naltrexone block
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: Oxycodone — 1X40 mg PF-00345439 formulation A capsule with water and under fed condition
  Arms: Oxycodone Formulation A Capsule
Drug: Oxycodone — 1X40 mg PF-00345439 formulation B capsule with water and under fed condition
  Arms: Oxycodone Formulation B Capsule
Drug: Oxycodone — 1X40 mg PF-00345439 formulation C capsule with water and under fed condition
  Arms: Oxycodone Formulation C Capsule
Drug: Oxycodone — 1X40 mg PF-00345439 formulation D capsule with water and under fed condition
  Arms: Oxycodone Formulation D Capsule
Drug: Oxycodone — 40 mg oxycodone oral solution (5 mg/5 ml) with water and under fed condition
  Arms: Oxycodone Oral Solution

SUMMARY:
To estimate the pharmacokinetics and relative bioavailability of oxycodone after administration of 40 mg doses of four PF-00345439 formulations and oxycodone in solution

DETAILED DESCRIPTION:
This study will estimate the PK and relative bioavailability of oxycodone following single oral 40-mg doses of 3 modified PF-00345439 Formulations B, C, and D compared with the reference Formulation A under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 21 and 55 years, inclusive

Exclusion Criteria:

* Evidence or history of clinically significant diseases

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) (if data permit, otherwise Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUClast]) of oxycodone. | 0, 0.5, 1, 2, 4, 6, 8, 12, 14, 16, 24, 36, 48 hours post-dose
Maximum Observed Plasma Concentration (Cmax) | 0, 0.5, 1, 2, 4, 6, 8, 12, 14, 16, 24, 36, 48 hours post-dose

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of oxycodone, as data permit. | 0, 0.5, 1, 2, 4, 6, 8, 12, 14, 16, 24, 36, 48 hours post-dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) of oxycodone, as data permit. | 0, 0.5, 1, 2, 4, 6, 8, 12, 14, 16, 24, 36, 48 hours post-dose
Plasma Decay Half-Life of oxycodone, as data permit. | 0, 0.5, 1, 2, 4, 6, 8, 12, 14, 16, 24, 36, 48 hours post-dose
Concentration at time 24 hours (C24) of oxycodone, as data permit. | 0, 0.5, 1, 2, 4, 6, 8, 12, 14, 16, 24, 36, 48 hours post-dose
Adverse events, vital signs and laboratory parameters. | 0, 0.5, 1, 2, 4, 6, 8, 12, 14, 16, 24, 36, 48 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4501010&StudyName=Pharmacokinetics%20And%20Relative%20Bioavailability%20Study%20Of%20Oxycodone%0A